CLINICAL TRIAL: NCT00560586
Title: Nasal Budesonide in Children With Rhinitis and/or Mild Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 388.03; UofL Project ID 04-0280X02
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep fragmentation; apnea; hypoxia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Deprivation; Apnea; Hypoxia | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Experimental): Budesonide for 6 weeks followed by crossover to placebo
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Placebo for 6 weeks followed by crossover to treatment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Budesonide — 1 puff each nostril (32 micrograms) at bedtime
  Arms: Budesonide
Drug: placebo — 1 puff each nostril at bedtime
  Arms: Placebo

SUMMARY:
-Intranasal budesonide therapy may lead to improved symptoms and sleep study findings in children with mild obstructive sleep apnea with and without allergic rhinitis that would not be treated with T&A. The aim of the study is to conduct a randomized double blind cross-over trial comparing the effect of once a day intranasal budesonide therapy vs. placebo in children with mild sleep apnea that would not be candidates for T&A.

DETAILED DESCRIPTION:
Untreated OSAS can result in serious morbidity, primarily affecting neurobehavioral and cardiovascular systems.

The severity of OSAS is only partially related to the adenoid and tonsillar size. While adenotonsillectomy (T&A) is the most common treatment for children with OSAS, this approach is reserved for children whose apnea/hypopnea index in the overnight sleep study exceeds a critical value. However, there is no consensus on the appropriate management of children with AHI >1 but <7 events/hour of sleep. These children constitute between 4-6% of all children and there are no alternative long-term interventions, and therefore a medical approach that obviates surgery, yet leads to substantial amelioration in the sleep-disordered breathing is critically needed.

Anti-inflammatory agents like intra-nasal corticosteroids are considered an effective treatment for children with allergic rhinitis. However, only one study has been conducted so far, and has examined the effect of intranasal corticosteroids, in pediatric patients with florid OSAS. Thus, no studies are available on topical steroids in patients with OSAS severity that would not justify T&A.

Our leading hypothesis is:

- Intranasal budesonide therapy may lead to improved symptoms and polysomnographic findings in children with OSAS with and without allergic rhinitis that would not be treated with T&A.

Subjects And Methods Study population Specific Aim. Up to 100 children will be recruited from all pediatric patients referred for evaluation of snoring and who underwent clinical evaluation, lateral neck x-ray, and an overnight sleep study at the Kosair Children's Hospital Sleep Medicine and Apnea Center.

Study Design Specific Aim: After informed consent is obtained from the parents, children fulfilling the entry criteria will be randomized using a table of random numbers that will be provided by Astra-Zeneca. Patients will be allocated into parallel treatment groups with simple randomization in blocks of 4 in a double blind fashion, according to the randomization procedure delineated by Astra-Zeneca All patients will complete a questionnaire regarding symptoms of snoring and allergic rhinitis symptoms prior to starting the study. One of the groups will start a-6 week course of either nasal topical budesonide (32 mcg/puff/nostril to both nostrils (total of 64 mcg), once a day or placebo. Parents will be instructed to give the drug at bedtime. Parents will be contacted weekly by the investigators to determine whether the study drug is being given as prescribed. When unable to contact parents by phone, they will be sent a follow up letter accompanied with the weekly questionnaire and a postage-paid return envelope. After 6 weeks, patients will have an overnight sleep study, lateral neck x-ray, and they will fill in a questionnaire regarding snoring and rhinitis symptoms.. At the end of the 6 weeks, patients will start a 6-week course with the compound that they were not receiving during the 1st phase of the study. All the outcome endpoints will be assessed again upon completion of the 2nd 6-week course.

The overall rationale for this schedule is as follows:

We are aiming to assess whether intranasal budesonide is effective in ameliorating sleep-disordered breathing in these children. Therefore, we aim to maximize the number of children receiving intranasal budesonide. This is achieved in the above experimental scheme since all children will receive 6 weeks of the therapy, either at the onset of their 12-week participation or after 6 weeks (for those who will be randomized to placebo treatment in the initial 6 weeks). The rationale for a 6-week duration period is that we anticipate that the reduction in adenoid volume will be a slow process that requires between 3-6 weeks to reach its peak effect. We also wish to determine whether cessation of intranasal budesonide is associated with exacerbation of the SDB. To this effect, the group of children who were initially treated with budesonide for 6 weeks will provide the data towards answering this important question. We anticipate that rebound increase in severity will occur but may take several weeks to manifest since the incremental growth of adenoid tissue will also take time.

Both nasal-budesonide and placebo inhalers will be provided in identical containers by the drug manufacturer. The appearance and smell of the budesonide and placebo will be indistinguishable. The investigators will not be aware of the compound being used. The codes for each patient will be kept by Astra-Zeneca. If any adverse event develops, the patients will be withdrawn from the study and followed clinically to assess overall clinical course.

Experimental Protocols

Symptoms questionnaire All patients will fill a snoring and symptom questionnaire.

Lateral Neck X-Rays This will be performed using standard techniques in the Radiology Department at KCH.

Overnight Polysomnography All children participating in the study will be polysomnographically studied before inclusion as part of their routine clinical evaluation. In addition, they will undergo 2 additional sleep studies, each at the end of the 6-week intervention period of the study.

Statistics A sample size of 50 patients per arm in this parallel design study was estimated based on an alpha error of 0.05, beta error of 0.2, a baseline mean apnea hypopnea index (AHI) of 3, with an SD of 1.5, and a potential decrease in AHI by 20%. In addition, such number of subjects would allow for detection of a 30% improvement in rhinitis scores. Even if attrition occurs, 40 subjects per arm will be sufficient assuming a 30% improvement in AHI according to sleep study. This design and number will also permit accurate determination of rebound exacerbation following transition from budesonide to placebo in half the subjects. (see above). Results will be expressed as the mean +/- SEM. To assess treatment effectiveness, paired t-tests will be used to compare normally distributed variables.

Potential Risks Nasal budesonide (Rhinocort Aqua, AstraZeneca) is generally well tolerated.. The most commonly reported adverse events( more then 2%) for Rhinocort Aqua and vehicle placebo (a formulation with no active drug) respectively were: epistaxis (nosebleed) - 8 percent vs 5 percent; pharyngitis (sore throat) - 4 percent vs 3 percent; bronchospasm 2 percent vs 1 percent; nasal irritation - 2 percent vs <1 percent; and coughing - 2 percent vs <1 percent.

Rare adverse events reported include: nasal septum perforation, pharynx disorders (throat irritation or pain, swollen throat, burning throat, itching throat, angioedema, anosmia and palpitations. Even though, studies have shown detectable adrenal suppression with intranasal steroids administration,30 intranasal budesonide 200 µg once daily has been found to have no effects on 24 hour, or fractionated cortisol profiles in serum or urine.31 And although transient growth suppression have been reported with medium to high dose inhaled steroids, no similar side effects were reported during clinical studies with intranasal budesonide. Furthermore, the addition of intranasal budesonide therapy to medium dose of inhaled budesonide in children with asthma for approximately 24 months had no significant effect on final adult height.32

Potential Benefits It is possible that the participants will have improvements in the severity of their OSAS and their snoring severity during nasal budesonide therapy.

The information obtained in our study, will help to define the role of nasal budesonide intervening in the pathophysiology of OSAS, and the potential role of nasal budesonide as a nonsurgical therapy for children with otherwise mild OSAS who would not be considered as candidates for T&A.

Significance of Research For children with OSAS that is too mild to justify T&A surgery, Intranasal therapy with budesonide may become a safe and effective new therapy aiming to minimize the morbidity associated with OSAS in children.

ELIGIBILITY:
Inclusion Criteria:

* Children >6 years of age and < 12 years of age, who snore and have an apnea hypopnea index (AHI) < or equal 7 or Respiratory arousal index > or equal 2

Exclusion Criteria:

* Hypersensitivity to budesonide
* Recent nasal trauma
* Nasal surgery or nasal septum perforation
* Current therapy with drugs interacting with budesonide (erythromycin clarythromycin, ketoconazole and cimetidine)
* Immunodeficiency or immunosuppressant therapy
* Craniofacial, neuromuscular, syndromic or defined genetic abnormalities
* Acute upper respiratory tract infection
* Systemic corticosteroid therapy or antibiotic therapy in the 2 weeks previous to the study, and
* Children who already had adenotonsillectomy in the past 12 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in the number of apnea/hypopnea episodes during a sleep study | Start of study, 6 weeks after drug treatment started and 6 weeks after placebo treatment started.
  Subjects will complete a sleep study with polysomnography at beginning of treatment and 6 weeks after start of treatment. Analysis of the sleep study will provide the number of times the subject has apnea (temporary cessation of breathing) or hypopnea (slow or shallow breathing)

SECONDARY OUTCOMES:
Pediatric sleep questionnaire (PSQ) at baseline | Start of study
  The PSQ is a 67 item instrument which has been validated in a wider age range, 4 to 18 years. The answers to the questions on the PSQ are: yes/no/don't know, which makes it simpler to use. The PSQ covers a wide range of sleep problems in children and has a sleepiness subscale, and a sleep related breathing disorder subscale, (which is the only non-PSG tool found to be useful in identifying obstructive sleep apnea). The PSQ has been used in clinical research and is applicable to screening as well. The scoring of this questionnaire will allow the investigators to determine any change in the quality of the subject's sleep.
Pediatric sleep questionnaire (PSQ) after treatment | 6 weeks after drug treatment started
  The PSQ is a 67 item instrument which has been validated in a wider age range, 4 to 18 years. The answers to the questions on the PSQ are: yes/no/don't know, which makes it simpler to use. The PSQ covers a wide range of sleep problems in children and has a sleepiness subscale, and a sleep related breathing disorder subscale, (which is the only non-PSG tool found to be useful in identifying obstructive sleep apnea). The PSQ has been used in clinical research and is applicable to screening as well. The scoring of this questionnaire will allow the investigators to determine any change in the quality of the subject's sleep.
Pediatric sleep questionnaire (PSQ) after placebo | 6 weeks after placebo treatment started.
  The PSQ is a 67 item instrument which has been validated in a wider age range, 4 to 18 years. The answers to the questions on the PSQ are: yes/no/don't know, which makes it simpler to use. The PSQ covers a wide range of sleep problems in children and has a sleepiness subscale, and a sleep related breathing disorder subscale, (which is the only non-PSG tool found to be useful in identifying obstructive sleep apnea). The PSQ has been used in clinical research and is applicable to screening as well. The scoring of this questionnaire will allow the investigators to determine any change in the quality of the subject's sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Leila Kheirandish, MD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital Sleep Center, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Kheirandish-Gozal L, Gozal D. Intranasal budesonide treatment for children with mild obstructive sleep apnea syndrome. Pediatrics. 2008 Jul;122(1):e149-55. doi: 10.1542/peds.2007-3398. PMID 18595959